CLINICAL TRIAL: NCT00789893
Title: A Descriptive Study of Vaginal Dilator Use After Pelvic Radiotherapy
Brief Title: Study of Vaginal Dilator Use After Pelvic Radiotherapy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-127
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Cancer; Endometrial Cancer; Rectal Cancer; Anal Cancer
Keywords: external beam pelvic radiation; brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Rectal Neoplasms; Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Women with cervical, endometrial, rectal or anal cancer: Women seen in the radiation oncology clinic with cervical, endometrial, rectal or anal cancer who will receive external beam pelvic radiation or brachytherapy
  Interventions: Device: Vaginal Dilator

INTERVENTIONS:
Device: Vaginal Dilator — Participants will be instructed to use the dilators 3 times per week, regardless of frequency of sexual intercourse. At 5 time points, data will be collected to determine vaginal dilator size, grade vaginal stenosis & assess vaginal symptoms. 1)Baseline: patient self-assessment following consultation up until the end of the first week of radiation 2)Post-radiation: patient self-assessment one month ± 2 weeks follow-up from last day of radiation 3)Post-radiation: 3 month ± 4 weeks follow-up from initiation of dilator use 4)Post-radiation: 6 month ± 4 weeks follow-up from initiation of dilator use 5)Post-radiation: 12 months ± 4 weeks follow-up from initiation of dilator use. At the 1st & 2nd time points, the nurse will telephone the patient to retrieve her responses. The 1st phone call will occur between the time following consultation up until the end of the first week of radiation, & the 2nd will be one month ± 2 weeks from last day of radiation.
  Other Names: The remaining assessments will be performed during the patient's regularly; scheduled follow-up appointments or via phone calls.

SUMMARY:
Patient will have radiation to treat the cancer. This treatment can make the vagina both narrower and shorter. That can cause two problems. It can make it harder for the doctor to do a pelvic exam during a follow-up visits. And, it can make sexual intercourse uncomfortable.

We tell women to use a vaginal dilator after radiation to the pelvis. This is standard education. We do not routinely ask women how they do with it. We are doing this study to see if using the dilator as we instruct will help the vagina stretch. The patient will have an examine of the vagina before the start of radiation. We will see what size dilator can fit. The goal of this study is to have the patient be able to use that size dilator within six months after radiation.

ELIGIBILITY:
Inclusion Criteria:

* Female with cervical, endometrial, rectal or anal cancer
* Scheduled to begin one of the following treatments at MSKCC:
* Definitive external beam radiation therapy
* Preoperative external beam radiation therapy of followed by surgery
* Postoperative external beam radiation therapy
* Definitive external beam radiation therapy with intracavitary brachytherapy (tandem and ring or Syed)± surgery
* Postoperative intravaginal brachytherapy (once every two weeks times three)
* ≥ or = to 21 years of age

Exclusion Criteria:

* Women with cervical, endometrial, rectal or anal cancer who are/have:
* Unable to speak and write English so that it would prohibit them from full participation in the study. Patient education, instruction and questionnaire are validated in English.
* Mental or physical handicaps that would prohibit them from full participation in the study.
* Prior radiation to the pelvis.
* Evidence of metastatic disease.

Ages: 21 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women seen in the radiation oncology clinic with cervical, endometrial, rectal or anal cancer who will receive external beam pelvic radiation or brachytherapy.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To measure compliance with vaginal dilator use. | conclusion of study
To examine the effect of dilator use in minimizing vaginal stenosis so that patients are able to use the pre-radiation baseline dilator size 6 months after starting dilator use. | conclusion of study

SECONDARY OUTCOMES:
To measure vaginal symptoms related to vaginal stenosis during vaginal dilation over 6 months after starting dilator use. | conclusion of study
To explore reasons for non-compliance with use of dilators. | conclusion of study
To explore patient-reported self-efficacy as it relates to the use of the vaginal dilator. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Ethel Law, MA, RN, OCN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org